CLINICAL TRIAL: NCT01245686
Title: A Combined Lifestyle and Medication Intervention to Reduce CVD Risk
Brief Title: Heart to Health: A Combined Lifestyle and Medication Intervention to Reduce Cardiovascular Disease (CVD) Risk
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Principal Investigator, Thomas Keyserling, MD, MPH, Professor of Medicine, University of North Carolina, Chapel Hill
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 10-2028; 1U48DP002658 (NIH)
Record Dates: First submitted 2010-11-19; First posted 2010-11-22 (Estimated); Last update posted 2013-02-06 (Estimated); Status verified 2013-02

CONDITIONS: Cardiovascular Disease; Coronary Heart Disease
Keywords: Diet interventions; Physical activity interventions; Medication adherence; Tailored interventions
MeSH Terms: conditions — Cardiovascular Diseases; Coronary Disease; Medication Adherence

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- One-on-one counseling (Active Comparator): Participants in this arm will receive 4 intensive one-on-one counseling sessions (either in person or on the phone) and 3 brief maintenance sessions.
  Interventions: Behavioral: Lifestyle and medication intervention
- Web counseling (Active Comparator): Participants in this arm will receive 4 intensive counseling sessions over the web. They will also receive 3 maintenance sessions over the web.
  Interventions: Behavioral: Lifestyle and medication intervention

INTERVENTIONS:
Behavioral: Lifestyle and medication intervention — The Heart to Health Intervention combines and enhances two previously tested interventions to reduce CVD risk (a counselor-based intervention to improve lifestyle and a web-based intervention to improve medication adherence). The new lifestyle and medication adherence intervention (delivered alternately in a one-on-one counseling or web-format) includes a decision aid on heart disease risk and risk-reducing options, general education on lifestyle and medication adherence, tips for overcoming barriers to CHD risk reduction, and goal setting and specification of first steps.

SUMMARY:
Cardiovascular disease (CVD), including heart disease and stroke, is the leading cause of death in the US. Every year, more than one million Americans have a heart attack, and nearly 800,000 have a stroke. In 2010, heart disease alone is expected to cost the country more than $316 billion in health care and lost productivity.

Both lifestyle changes and medication can reduce the risk of CVD, and this project combines these approaches in the hopes of identifying a practical intervention for use in primary care medical offices. The project combines two previously tested interventions and updates them to meet current guidelines for diet and use of aspirin and cholesterol-controlling drugs (statins).

The research team is delivering the combined intervention in two formats: web-based and counselor-based. Each format has the same content, but the web-based advice is accessed through the Internet by clients at home, a community site, or a primary care office. The other format involves sessions delivered to clients by a counselor either in person at a primary care office or over the telephone. The researchers will compare how effective each format is in reducing participants' risk of coronary heart disease. They will also determine the interventions' effect on participants' diet, physical activity, smoking status, medication adherence, and other health indicators. In addition, the team will compare the two formats' cost-effectiveness and how well the patients, office staff, and clinicians accept the interventions.

Recruited from five family practices, 600 patients representing the geographic and ethnic diversity of North Carolina are taking part in this study. Half the participants are randomly assigned to the web-based intervention; the other half to the counselor-based version. Both groups will also get information on local resources, such as gyms and farmers markets, that can help participants maintain a healthy lifestyle.

ELIGIBILITY:
Inclusion Criteria:

* Established patients
* Men ages 35-79
* Women ages 45-79
* History of CVD (100 participants)
* CHD risk equal or greater than 10%
* elevated CHD risk factor

Exclusion Criteria:

* non-English speaking
* no phone
* treatment of psychosis
* history of alcohol/substance abuse within last 2 years
* pregnancy, breast feeding, or anticipated pregnancy in next 18 months
* history of malignancy, other than non-melanoma skin cancer, that has not been in remission or cured surgically for >5 years
* recent history (in past year) of hypoglycemic event requiring medical attention
* estimated creatinine clearance less than 30 ml/min

Ages: 35 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 489 (Actual)
Dates: Start 2011-02; Primary Completion 2012-07 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Predicted 10-year CHD risk | 4-month follow-up
  Framingham risk scores are well-validated and provide an absolute estimate of the likelihood of CHD events (MI, angina, and CHD death) over a 10-year time period.
  We will examine absolute changes in this outcome in both intervention arms. We will also examine whether this outcome varies by subgroups of the following variables: baseline level of predicted CHD risk, age, race, SES, insurance status, overall health status, numeracy, literacy, # medications, # of perceived barriers to adherence, use of the intervention, time with the intervention, study practice site, and health counselor

SECONDARY OUTCOMES:
Predicted 10-year CHD risk | 12 months
  Framingham risk scores are well-validated and provide an absolute estimate of the likelihood of CHD events (MI, angina, and CHD death) over a 10-year time period.
Use of and adherence to cardiovascular medicines | 4 and 12 months
  Use of cardiovascular medicines will be by self-report. Adherence to cardiovascular medicines will be measured by the 8-Item Morisky scale and a single-item specifying overall percentage adherence to cardiovascular medicines(categorical).
  Participants will additionally report use of and adherence to individual medicines, including aspirin, blood pressure medicine, and cholesterol medicine. Aspirin adherence will be validated by serum thromboxane b2 in a subsample of participants. Blood pressure and cholesterol medicine use will be confirmed by changes in blood pressure and cholesterol.
Dietary Intake | 4 and 12 months
  Dietary intake will be measured through a combination of self-report and objective measures. Participants will self-report diet on two validated questionnaires: the block questionnaire (fruit and vegetable intake) and the fat quality screener. Fruit and vegetable intake will be objectively measured by serum carotenoids. Fat quality will be objectively measured using RBC membrane fatty acids.
Physical activity | 4 and 12 months
  Physical activity will be measured through a combination of self-report and objective measures. Participants will report physical activity on the validated modified RESIDE questionnaire. They will additionally wear a pedometer to monitor their daily total and aerobic steps.
Blood pressure | 4 and 12 months
  Blood pressure will be measure via standardized protocol using an oscillometric automatic monitor
Total, HDL, and direct LDL cholesterol | 4 and 12 months
  Total, HDL, and direct LDL cholesterol will be measured via enzymatic calorametric testing.
Smoking status | 4 and 12 months
  Smoking will be measured through a combination of self-report and urinary cotinine (Nicalert test strips).
Adverse events | 4 and 12 months
  We will monitor the following adverse events: ED visits (self-report), hospitalizations (self-report), deaths (family report confirmed by death registry), GI bleeds (self-report), hemorrhagic stroke (self-report), musculoskeletal injury (self-report), renal dysfunction (serum creatinine), and liver dysfunction (AST).
Acceptability of the Intervention | 4 and 12 months
  We will measure the acceptability of the intervention using process measures querying participants, office staff, and clinicians about the perceptions of the acceptability of the intervention and the time to deliver it.
Cost-effectiveness | 4 and 12 months
  We will measure the cost-unit CHD risk reduction for the two interventions using a societal perspective.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas C Keyserling, MD, MPH, Principal Investigator — UNC-Chapel Hill; Stacey L Sheridan, MD, MPH, Study Director — UNC-Chapel Hill
Locations (5):
- United States (5):
  - Durham Family Practice, Durham, North Carolina
  - Dayspring Family Medicine, Eden, North Carolina
  - Cabarrus Family Medicine Residency, Kannapolis, North Carolina
  - Moncure Community Health Center, Moncure, North Carolina
  - Caswell Family Medical Clinic, Yanceyville, North Carolina

REFERENCES:
- [Derived] Keyserling TC, Sheridan SL, Draeger LB, Finkelstein EA, Gizlice Z, Kruger E, Johnston LF, Sloane PD, Samuel-Hodge C, Evenson KR, Gross MD, Donahue KE, Pignone MP, Vu MB, Steinbacher EA, Weiner BJ, Bangdiwala SI, Ammerman AS. A comparison of live counseling with a web-based lifestyle and medication intervention to reduce coronary heart disease risk: a randomized clinical trial. JAMA Intern Med. 2014 Jul;174(7):1144-57. doi: 10.1001/jamainternmed.2014.1984. PMID 24861959
- [Derived] Sheridan SL, Draeger LB, Pignone MP, Sloane PD, Samuel-Hodge C, Finkelstein EA, Gizlice Z, Vu MB, Gitterman DP, Bangdiwala SI, Donahue KE, Evenson K, Ammerman AS, Keyserling TC. Designing and implementing a comparative effectiveness study of two strategies for delivering high quality CHD prevention: methods and participant characteristics for the Heart to Health study. Contemp Clin Trials. 2013 Nov;36(2):394-405. doi: 10.1016/j.cct.2013.07.013. Epub 2013 Aug 2. PMID 23916919